CLINICAL TRIAL: NCT04925037
Title: Explore the Associations of Behavioral Factors With Treatment Adherence in Axial Spondyloarthritis Patients Treated With Biotherapy
Acronym: MAINTAIN II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 TOURNADRE
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Axial Spondyloarthritis
Keywords: Adherence; Biologic treatment; Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: self-questionnaire to patients undergoing SpAax follow-up — On the occasion of a single visit in consultation or hospitalization, an anonymous self-questionnaire will be distributed to patients undergoing SpAax follow-up

SUMMARY:
The management of chronic inflammatory rheumatism, including spondyloarthritis (SpA), has been revolutionized in recent decades with the arrival of biological therapy. The success of the current therapeutic strategy is also based on therapeutic compliance. If therapeutic adherence in rheumatoid arthritis patient (RA) is only 66%, it seems even worse in SpA. Few studies report quantitatively the adherence of SpA patients, as well as the predictive or associated factors. The objective of this study is to assess the patient adherence to biologics in patients with axial SpA (SpAax), and to investigate factors influencing this adherence, in particular the association with vaccination coverage, dietary behavior, and digital health tools.

DETAILED DESCRIPTION:
Multicentric cross-sectional survey of patients seen in the context of a rheumatology consultation or hospitalization.

On the occasion of a single visit in consultation or hospitalization, an anonymous self-questionnaire will be distributed to patients undergoing SpAax follow-up to assess their compliance with biologic drugs, their vaccination coverage, their diet, the presence of a fibromyalgia syndrome or inflammatory bowel disease, intestinal disorders, regular physical activity and sedentary lifestyle, the frequency and mode of use of mobile applications and/or connected objects related to health, the presence of catastrophic thoughts and the presence of anxiety and depressive disorders. Medical data relevant to routine care will be collected.(Age, sex, weight, height, tobacco and alcohol use, disease characteristics, SpA treatment, comorbidities)

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years old with axial spondyloarthritis according to ASAS criteria and treated with biotherapy.
* French-speaking, without any understanding problems.

Exclusion Criteria:

* Patients under curatorship, guardianship or other legal protection
* Patients refusing to consent to participate in research
* Pregnant and breastfeeding women.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with axial spondyloarthritis according to ASAS criteria and treated with biotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-06-21 (Estimated); Study Completion 2022-06-21 (Estimated)

PRIMARY OUTCOMES:
adherence to biotherapies | Day 1
  Proportion of spondyloarthritis patients with good adherence to biotherapies. Adherence was assessed by Girerd's self-administered questionnaire score.
  Six questions self-questionnaire, Yes =1 and No = 0
  Patients are then classified as follows:
  * Score = 0: Good adherence to therapy
  * Score = 1 or 2: minimal adherence problem
  * Score > 3: Poor adherence to therapy

SECONDARY OUTCOMES:
Proportion of patients who received influenza and pneumococcal vaccinations | Day 1
  The patient checks on the self-questionnaire if he is vaccinated or not against influenza and pneumococcus
Proportion of vaccinated patients with good adherence to biologic treatment. | Day 1
  Proportion of patients who indicated to be vaccinated and who has a GIRERD score =0
Proportion of patients using digital health tools with good adherence to biologic treatment. | Day 1
  Proportion of patients who checked yes for users of digital health tools with a GIRERD score =0
Proportion of patients on a diet and good adherence to biologic treatment. | Day 1
  Proportion of patients who reported being on a diet with a GIRERD score = 0
Proportion of Inflammatory bowel disease (IBD) patients with good adherence to biologic treatment | Day 1
  Proportion of patients with crohn's disease or ulcerative colitis indicated by the physician with a GIRERD score =0
Proportion of patients with regular physical activity and good adherence to biologic treatment. | Day 1
  Proportion of patients who are physically active every day (defined by the World Health Organisation as 150 minutes per week of moderate intensity activity, or 75 minutes of high intensity activity ) and have a GIRERD score =0
Proportion of fibromyalgia patients with good adherence to biologic treatment | Day 1
  Fibromyalgia diagnosis will be evaluated by the answers to the Fibromyalgia Rapid Screening Tool self-questionnaire. 6-question closed-ended questionnaire. (YES=1, NO=0). Score ≥ 5 = Fibromyalgia confirmed.
  Proportion of patient who have a score GIRERD = 0 and FiRST score ≥ 5
Proportions of patients with catastrophic thoughts and good adherence to biologic treatment. | Day 1
  the Patient Catastrophing Scale (PCS) is a broad self report measure of pain catastrophizing and consists of 13 items scored using a 5-point Likert scales from 0 (never) to 4 (always) points. The total score for the PCS equals 52. Responses are summed to create a total score, with higher scores indicating greater pain catastrophizing levels. A score of more than 24 indicates a high level of catastrophizing.
Proportions of patients with anxiety and depressive disorders in patients with good adherence to biologic treatment | Day 1
  Anxiety and depression disorders were assessed by the Hospital Anxiety and Depression Scale (HADS). The HADS questionnaire is composed of two parts: one part includes 7 items for screening for depression; and a second one also includes 7 items for the screening for anxiety disorders. A score between 0 and 3 is assigned to each item. The score total per party varies between 0 and 21. Score ≥ 11 = Anxiety or depression confirmed.
  Proportion of patient who has HADS-anxiety and/or HADS-depression ≥ 11 and a GIRERD score = 0.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Bordeaux, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Limoges, Limoges
  - CHU Montpellier, Montpellier
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No